CLINICAL TRIAL: NCT00642460
Title: A Randomized, Placebo-controlled Study to Evaluate the Effect of Tocilizumab on Disease Response in Patients With Active Systemic Juvenile Idiopathic Arthritis (JIA), With an Open-label Extension to Examine the Long Term Use of Tocilizumab
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Patients With Active Systemic Juvenile Idiopathic Arthritis (JIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WA18221; 2007-000872-18
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab; Anti-Inflammatory Agents, Non-Steroidal; Methotrexate; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: Non-steroidal anti-inflammatory drugs (NSAIDs); Drug: methotrexate; Drug: corticosteroids
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Non-steroidal anti-inflammatory drugs (NSAIDs); Drug: methotrexate; Drug: corticosteroids

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg (patients>=30kg) or 12mg/kg (patients <30kg) iv every 2 weeks. In Part III, administration frequency may be reduced to every 3 and every 4 weeks, respectively, according to an optional alternative dosing schedule.
  Arms: 1
Drug: Placebo — iv every 2 weeks for 12 weeks
  Arms: 2
Drug: Non-steroidal anti-inflammatory drugs (NSAIDs) — as prescribed
Drug: methotrexate — as prescribed
Drug: corticosteroids — orally, as prescribed

SUMMARY:
This study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in patients with active systemic juvenile idiopathic arthritis (sJIA) who have an inadequate clinical response to NSAIDs and corticosteroids. In Part I of the study patients will be randomized 2:1 to receive iv infusions of RoActemra/Actemra (8mg/kg iv for patients >=30kg, or 12mg/kg for patients <30kg) or placebo, every 2 weeks. Stable NSAIDs and methotrexate will be continued throughout. After 12 weeks of double-blind treatment, all patients will have the option to enter Part II of the study to receive open-label treatment with RoActemra/Actemra for a further 92 weeks, followed by a 3-year continuation of the study in Part III in which, for patients who meet specific criteria, an optional alternative dosing schedule decreasing the study drug administration frequency will be introduced. Anticipated time on study treatment is up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2-17 years of age
* Systemic juvenile idiopathic arthritis with >= 6 months persistent activity
* Presence of active disease (>=5 active joints, or >=2 active joints + fever + steroids)
* Inadequate clinical response to nonsteroidal anti-inflammatory drugs (NSAIDs) and corticosteroids due to toxicity or lack of efficacy

Exclusion Criteria:

* Wheelchair-bound or bed-ridden
* Any other autoimmune, rheumatic disease or overlap syndrome other than systemic juvenile idiopathic arthritis
* Intravenous long-acting corticosteroids or intra-articular corticosteroids within 4 weeks of baseline, or throughout study
* Disease-modifying antirheumatic drugs (DMARDs), other than methotrexate
* Previous treatment with tocilizumab

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (13):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Hartford, Connecticut
  - Augusta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Hackensack, New Jersey
  - Livingston, New Jersey
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas
- Argentina (2):
  - Buenos Aires
  - La Plata
- Australia (3):
  - Parkville
  - Subiaco
  - Westmead
- Belgium (2):
  - Ghent
  - Leuven
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (4):
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Ottawa, Ontario
  - Toronto, Ontario
- Prague, Czechia
- Copenhagen, Denmark
- Germany (3):
  - Berlin
  - Bremen
  - Sankt Augustin
- Greece (3):
  - Athens
  - Heraklion
  - Ioannina
- Italy (4):
  - Genova
  - Milan
  - Padua
  - Roma
- Mexico (2):
  - México
  - Miexico City
- Utrecht, Netherlands
- Oslo, Norway
- Poland (2):
  - Krakow
  - Lublin
- Piešťany, Slovakia
- Spain (4):
  - Barcelona
  - Esplugas de Llobregat
  - Madrid
  - Valencia
- Gothenburg, Sweden
- United Kingdom (2):
  - Liverpool
  - London

REFERENCES:
- [Derived] Malattia C, Ruperto N, Pederzoli S, Palmisani E, Pistorio A, Wouters C, Dolezalova P, Flato B, Garay S, Giancane G, Wells C, Douglass W, Brunner HI, De Benedetti F, Ravelli A; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Tocilizumab may slow radiographic progression in patients with systemic or polyarticular-course juvenile idiopathic arthritis: post hoc radiographic analysis from two randomized controlled trials. Arthritis Res Ther. 2020 Sep 10;22(1):211. doi: 10.1186/s13075-020-02303-y. PMID 32912276
- [Derived] Pardeo M, Wang J, Ruperto N, Alexeeva E, Chasnyk V, Schneider R, Horneff G, Huppertz HI, Minden K, Onel K, Zemel L, Martin A, Kone-Paut I, Siamopoulou-Mavridou A, Silva CA, Porter-Brown B, Bharucha KN, Brunner HI, De Benedetti F; Paediatric Rheumatology International Trials Organisation (PRINTO) and the Pediatric Rheumatology Collaborative Study Group (PRCSG). Neutropenia During Tocilizumab Treatment Is Not Associated with Infection Risk in Systemic or Polyarticular-course Juvenile Idiopathic Arthritis. J Rheumatol. 2019 Sep;46(9):1117-1126. doi: 10.3899/jrheum.180795. Epub 2019 Mar 1. PMID 30824645
- [Derived] De Benedetti F, Brunner H, Ruperto N, Schneider R, Xavier R, Allen R, Brown DE, Chaitow J, Pardeo M, Espada G, Gerloni V, Myones BL, Frane JW, Wang J, Lipman TH, Bharucha KN, Martini A, Lovell D; Paediatric Rheumatology International Trials Organisation and the Pediatric Rheumatology Collaborative Study Group. Catch-up growth during tocilizumab therapy for systemic juvenile idiopathic arthritis: results from a phase III trial. Arthritis Rheumatol. 2015 Mar;67(3):840-8. doi: 10.1002/art.38984. PMID 25504861
- [Derived] De Benedetti F, Brunner HI, Ruperto N, Kenwright A, Wright S, Calvo I, Cuttica R, Ravelli A, Schneider R, Woo P, Wouters C, Xavier R, Zemel L, Baildam E, Burgos-Vargas R, Dolezalova P, Garay SM, Merino R, Joos R, Grom A, Wulffraat N, Zuber Z, Zulian F, Lovell D, Martini A; PRINTO; PRCSG. Randomized trial of tocilizumab in systemic juvenile idiopathic arthritis. N Engl J Med. 2012 Dec 20;367(25):2385-95. doi: 10.1056/NEJMoa1112802. PMID 23252525

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of 3 parts. Part I: a 12 week double-blind placebo controlled study followed by Part II: a 92 week single arm open-label extension study followed by Part III: a 3 year open label continuation study.
Groups:
- Tocilizumab_8 mg/kg: Tocilizumab 8 mg/kg (for patients ≥30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part I and every 2 weeks for 92 weeks in Part II.
  Participants remained on their prescribed standard of care treatment with non-steroidal anti-inflammatory drugs (NSAIDs), methotrexate and corticosteroids if applicable.
- Tocilizumab_12 mg/kg: Tocilizumab 12 mg/kg (for patients <30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part I and every 2 weeks for 92 weeks in Part II.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
- Placebo: Placebo iv every 2 weeks for 12 weeks in Part 1. Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
- Tocilizumab Switchers: Tocilizumab Switchers includes all participants who changed their dose either Tocilizumab 8 mg/kg or 12 mg/kg intravenous (iv) every 2 weeks in Part II.
  Participants remained on their prescribed standard of care treatment with non-steroidal anti-inflammatory drugs (NSAIDs), methotrexate and corticosteroids if applicable.
- Participants ≥30 kg: Tocilizumab 8 mg/kg iv every 2 weeks for 12 weeks in Part I, every 2 weeks for 92 weeks in Part II and every 2 weeks for 156 weeks in Part III.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
- Participants <30 kg: Tocilizumab 12 mg/kg iv every 2 weeks for 12 weeks in Part I, every 2 weeks for 92 weeks in Part II and every 2 weeks for 156 weeks in Part III.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
Period: Part I: 12 Week Double-Blind
Arm/Group | Tocilizumab_8 mg/kg | Tocilizumab_12 mg/kg | Placebo | Tocilizumab Switchers | Participants ≥30 kg | Participants <30 kg
Started | 37 | 38 | 37 | 0 | 0 | 0
Part I : Intent-to-treat | 37 | 38 | 37 | 0 | 0 | 0
Completed | 36 | 37 | 36 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Refused Treatment | 1 | 0 | 0 | 0 | 0 | 0
Period: Part II: Open-Label Up to Week 92
Arm/Group | Tocilizumab_8 mg/kg | Tocilizumab_12 mg/kg | Placebo | Tocilizumab Switchers | Participants ≥30 kg | Participants <30 kg
Started | 52 (Includes Participants who received Open-Label in Part II or Open-Label escape therapy in Part I.) | 40 | 0 (Placebo group received open-label Tocilizumab 8 mg/kg or 12 mg/kg based on body weight in Part II.) | 20 (19 Participants switched from 12 mg/kg to 8 mg/kg and 1 Participant switched from 8mg/kg to 12 mg/kg) | 0 | 0
Part II: Intent-to-treat | 52 | 40 | 0 | 20 | 0 | 0
Completed | 43 | 32 | 0 | 17 | 0 | 0
Not Completed | 9 | 8 | 0 | 3 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Insufficient therapeutic response | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Refused treatment | 3 | 1 | 0 | 0 | 0 | 0
Not completed — Failure to return | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative reasons | 0 | 0 | 0 | 1 | 0 | 0
Period: Part III: Open-Label Up to Week 260
Arm/Group | Tocilizumab_8 mg/kg | Tocilizumab_12 mg/kg | Placebo | Tocilizumab Switchers | Participants ≥30 kg | Participants <30 kg
Started | 0 | 0 | 0 | 0 | 53 | 59
Completed | 0 | 0 | 0 | 0 | 28 | 38
Not Completed | 0 | 0 | 0 | 0 | 25 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 7 | 6
Not completed — Insufficient therapeutic response | 0 | 0 | 0 | 0 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Administrative reason | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused treatment | 0 | 0 | 0 | 0 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg (for patients ≥30 kg) or 12 mg/kg (for patients <30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part 1.
  Participants remained on their prescribed standard of care treatment with non-steroidal anti-inflammatory drugs (NSAIDs), methotrexate and corticosteroids if applicable.
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 75 | 37 | 112
Age, Customized [Number; unit: years]
  2 to 5 | 16 | 11 | 27
  6 to 12 | 33 | 15 | 48
  13 to 17 | 26 | 11 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 17 | 56
  Male | 36 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Part I: Percentage of Participants With ≥30% Improvement in Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) Core Set and Absence of Fever
Description: Percentage of participants with ≥30% improvement in ACR core set consisting of 6 components: 1) Physician's global assessment of disease activity Visual Analog Scale (VAS), 2) Parent/Patient global assessment of overall well-being VAS, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate, and 6) Childhood Health Assessment Questionnaire- Disability Index (CHAQ-DI) consisting of 30 questions in 8 domains.
  Absence of fever was defined as no diary temperature recording ≥37.5° Celsius in the preceding seven days.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population includes all participants who had at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg (for patients ≥30 kg) or 12 mg/kg (for patients <30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part 1.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 75 | 37
Percentage of participants | 85.3 | 24.3

2. Primary Outcome: Part II: Percentage of Participants With Decreases in Oral Corticosteroid Dose at Week 104
Description: Percentage of participants with ≥20 percent, ≥50 percent, ≥75 percent and ≥90 percent decreases in oral corticosteroid dose (mg/kg/day) from baseline.
Time Frame: Baseline, Week 104
Population: Includes only participants on oral corticosteroids at baseline.
Measure: Number; unit: Percentage of participants
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg (for patients >=30 kg) or 12 mg/kg (for patients <30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part 1.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 55
Percentage of participants
  ≥20 percent decrease | 76
  ≥50 percent decrease | 73
  ≥75 percent decrease | 62
  ≥90 percent decrease | 47

3. Secondary Outcome: Part I: Percentage of Participants With JIA Core Set ACR 30/50/70/90 Response at Week 12
Description: The six JIA ACR components consist of: 1) Physician's global assessment of disease activity, 2) Parent/Patient global assessment of overall well-being, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate, and 6) CHAQ-DI.
  At an assessment visit a JIA ACR30/50/70/90 response in comparison to Baseline is defined as: At least three of the six JIA ACR core components improving by at least 30%/50%/70%/90% and no more than one of the remaining JIA ACR core components worsening by more than 30%.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population includes all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 75 | 37
Percentage of participants
  JIA ACR30 response | 90.7 | 24.3
  JIA ACR50 response | 85.3 | 10.8
  JIA ACR70 response | 70.7 | 8.1
  JIA ACR90 response | 37.3 | 5.4

4. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Physician's Global Assessment of Disease Activity
Description: Physician's Global Assessment of disease activity is a Visual Analog Scale. The scale is 0 to 100 mm horizontal scale, the extreme left end of the line represents 'arthritis inactive' (i.e. symptom-free and no arthritis symptoms) and the extreme right end represents 'arthritis very active'. This item is completed by the treating physician.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are excluded. Last observation carried forward (LOCF) rule applied to missing JIA ACR core set components at Week 12.
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 73 | 17
Percentage change | -69.6 | -41.1

5. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Parent/Patient Global Assessment of Overall Well-being
Description: The Parent/Patient global assessment of overall well-being is a VAS. The scale is a 0 to 100 mm horizontal scale, the extreme left end of the line represents 'very well' (i.e. symptom-free and no arthritis disease activity) and the extreme right end represents 'very poor' (i.e. maximum arthritis disease activity). This item is completed by the patient or parent/guardian as appropriate.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are excluded. LOCF rule applied to missing JIA ACR core set components at Week 12.
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 73 | 17
Percentage change | -65.8 | -1.4

6. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Maximum Number of Joints With Active Arthritis
Description: The maximum number of joints with active arthritis is 71 and these are defined as those in the joint assessment with: swelling present or pain present and limitation of motion.
  The joint assessment is performed by an independent assessor, who is not the treating physician, blinded to all other aspects of the patient's efficacy and safety data.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 73 | 17
Percentage change | -70.6 | -37.2

7. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Number of Joints With Limitation of Movement
Description: The maximum number of joints with limitation of movement is 67 and these are defined as those in the joint assessment with 'limitation of motion'.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 72 | 17
Percentage change | -51.6 | -22.5

8. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Erythrocyte Sedimentation Rate
Description: Erythrocyte Sedimentation Rate (ESR) is an acute phase reactant measured in mm/hour.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 73 | 17
Percentage change | -88.2 | 33.6

9. Secondary Outcome: Part I: Percentage Change From Baseline in JIA Core Set ACR Score Component: Childhood Health Assessment Questionnaire Disability Index (CHAQ-DI)
Description: Functional ability is assessed using the CHAQ-DI. The questionnaire consists of 30 questions referring to eight domains; dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. Each domain has at least two component questions and if applicable to the patient there are four possible responses (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do).
  The CHAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score. This overall score ranges from 0 (best) to 3 (worst).
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Number; unit: Percentage change
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 72 | 17
Percentage change | -45.6 | -10.3

10. Secondary Outcome: Part I: Percentage of Participants With Fever Due to Systemic Juvenile Idiopathic Arthritis (sJIA) at Baseline Who Are Free of Fever at Week 12
Description: Fever free was defined as no diary temperature recording ≥37.5° Celsius in the preceding fourteen days.
Time Frame: Baseline, Week 12
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) who had a fever due to Systemic Juvenile Idiopathic Arthritis at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 41 | 24
Percentage of participants | 85.4 | 20.8

11. Secondary Outcome: Part I: Percentage of Participants With Changes in Laboratory Indicators: High-sensitivity C-Reactive Protein(hsCRP), Hemoglobin (Hb), Platelets and Leukocytes From Abnormal at Baseline to Normal at Week 12
Description: Percentage of participants with a change from an elevated hsCRP value at baseline to a normal hsCRP value at week 12; a change from anemia (low Hemoglobin) at baseline to a normal hemoglobin value at week 12; a change from thrombocytosis (elevated platelets) at baseline to a normal platelet value at week 12; a change from leukocytosis (elevated white blood cell count) at baseline to a normal white blood cell count at week 12.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population includes all randomized participants who received at least one dose of study drug. 'n' in each of the categories is the number of participants with data available at baseline and week 12 for analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 75 | 37
Percentage of participants
  hsC-Reactive Protein (n=72,34) | 98.6 | 5.9
  Hemoglobin (n=50,29) | 80.0 | 6.9
  Platelets (n=52,26) | 90.4 | 3.8
  Leukocytes (n=28,21) | 75.0 | 9.5

12. Secondary Outcome: Part I: Percentage of Participants With Concomitant Corticosteroid Reduction
Description: The percentage of participants receiving oral corticosteroids(CS) with a JIA ACR70 response at week 6 or Week 8 who reduced their oral CS dose by at least 20% without subsequent JIA ACR30 flare or occurrence of systemic symptoms at week 12.
  At an assessment visit a JIA ACR70 response is defined as: At least three of the six JIA ACR core components improving by at least 70% and no more than one of the remaining JIA ACR core components worsening by more than 30%.
Time Frame: Week 6 or Week 8, Week 12
Population: Participants from the Intent-to-treat population (all randomized participants who received at least one dose of study drug) who were taking oral corticosteroids.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 70 | 31
Percentage of participants | 24.3 | 3.2

13. Secondary Outcome: Part I: Change From Baseline in the Pain Visual Analog Scale (VAS) at Week 12
Description: Participants rated their pain by placing a horizontal line on a Visual Analog Scale on a scale of 0 (no pain)- 100 mm (severe pain). The score at 12 weeks minus the score at baseline. A negative number indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Intent-to-treat population who had Pain VAS data available at baseline and week 12. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are excluded. LOCF rule applied to missing pain VAS at Week 12.
Measure: Number; unit: mm
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 73 | 17
mm | -41.0 | -1.1

14. Secondary Outcome: Part I: Percentage of Patients With Minimally Important Improvement in CHAQ-DI Score at Week 12
Description: Percentage of patients who had at least a 0.13 improvement in CHAQ-DI score from Baseline to Week 12.
  The CHAQ-DI questionnaire consists of 30 questions referring to eight domains; dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. Each domain has at least two component questions and if applicable to the patient there are four possible responses (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do).
Time Frame: Baseline, Week 12
Population: Intent-to-treat Population. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are classified as non-responders.
  LOCF rule applied to missing CHAQ-DI Scores at Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 75 | 37
Percentage of participants | 77.3 [67.9 to 86.8] | 18.9 [6.3 to 31.5]

15. Secondary Outcome: Part I: Percentage of Patients With Rash at Baseline Who Are Free From Rash at Week 12
Description: Percentage of participants who had a rash characteristic of sJIA in the 14 days prior to the baseline visit but no rash characteristic of sJIA in the 14 days preceding the Week 12 visit day.
Time Frame: Baseline, Week 12
Population: Participants from the Intent-to-treat population for whom data was available. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are classified as non-responders.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 22 | 18
Percentage of participants | 63.6 [43.5 to 83.7] | 11.1 [0.0 to 25.6]

16. Secondary Outcome: Part I: Percentage of Patients With Anemia at Baseline With a ≥10 g/L Increase in Hemoglobin at Week 6 and Week 12
Description: Part I: Percentage of patients who had anemia (hemoglobin <lower level normal based on sex and age) at Baseline and a ≥10 g/L increase in hemoglobin at Week 6 and at Week 12.
Time Frame: Baseline, Week 6 and Week 12
Population: Participants from the Intent-to-treat population for whom hemoglobin data available. Patients who withdrew, received escape medication, or for whom the endpoint cannot be determined are classified as non-responders.
  LOCF rule applied to missing hemoglobin values at Week 6 and Week 12.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 50 | 29
Percentage of participants
  Week 6 | 88.0 [79.0 to 97.0] | 3.4 [0.0 to 10.1]
  Week 12 | 88.0 [79.0 to 97.0] | 3.4 [0.0 to 10.1]

17. Secondary Outcome: Part II: Percentage of Participants With JIA ACR70 and JIA ACR90 Responses Week 104
Description: The six JIA ACR components consist of: 1)Physician's global assessment of disease activity, 2)Parent/Patient global assessment of overall well-being, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate, and 6) CHAQ-DI.
  At an assessment visit a JIA ACR70/90 response in comparison to Baseline is defined as: At least three of the six JIA ACR core components improving by at least 70%/90% and no more than one of the remaining JIA ACR core components worsening by more than 30%.
Time Frame: Baseline, Week 104
Population: Participants from the Intent to Treat population who reached the time point plus patients who withdrew because of insufficient therapeutic response and are assumed to have been non-responders.
Measure: Number; unit: Percentage of Participants
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg (for patients >=30 kg) or 12 mg/kg (for patients <30 kg) intravenous (iv) every 2 weeks for 12 weeks in Part 1 and every 2 weeks for 92 weeks in Part II.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 75
Percentage of Participants
  JIA ACR70 response | 76.0
  JIA ACR90 response | 61.3

18. Secondary Outcome: Part II: Number of Active Joints at Week 104
Description: Seventy-one joints were assessed for signs of active arthritis. The mean number of joints with signs of active arthritis is reported.
Time Frame: Week 104
Population: Participants from the Intent to Treat population who reached this time point. No data imputation is applied and patients with missing data are excluded.
Measure: Mean (Standard Deviation); unit: Active Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 59
Active Joints | 1.9 (3.6)

19. Secondary Outcome: Part II: Percentage of Participants With no Active Joints at Week 104
Description: Seventy-one joints were assessed for signs of active arthritis. The percentage of participants with no signs of active arthritis is reported.
Time Frame: Week 104
Population: The Intent to Treat population in Part II includes 112 participants who received at least one dose of study drug. Only those participants who reached this time point are included in the analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 76
Percentage of Participants | 47.4

20. Secondary Outcome: Part II: Percentage of Participants With Inactive Disease at Week 104
Description: Criteria for Inactive Disease:
  1) No joints with active arthritis, 2) No fever, rash, serositis, splenomegaly, hepatomegaly (by physical exam) or generalized lymphadenopathy attributable to systemic juvenile idiopathic arthritis (sJIA), 3) Normal Erythrocyte Sedimentation Rate (<20 mm/hour), 4) Physician's global assessment of disease activity Visual Analog Scale (VAS) indicates no disease activity (where no disease activity is considered to be a score ≤10 mm on a 100 mm VAS).
Time Frame: Week 104
Population: Participants from the Intent to Treat population who reached time point plus patients who withdrew because of insufficient therapeutic response and are assumed to have been nonresponders.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 75
Percentage of Participants | 26.7

21. Secondary Outcome: Part II: Childhood Health Assessment Questionnaire-Disability Index (CHAQ-DI) Score at Week 104
Description: as for outcome 9
Time Frame: Baseline, Week 104
Population: Participants from the Intent to Treat population who withdrew have been excluded at post withdrawal visits.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 112
Score on a scale
  Baseline (n=112) | 1.68 (0.86)
  Week 104 (n=57) | 0.55 (0.71)

22. Secondary Outcome: Part II: Percentage of Participants With Oral Corticosteroid Cessation at Week 104
Description: Percentage is based on only those participants who were on oral corticosteroid at baseline and reached a nominal visit day on which dose was calculated.
Time Frame: Baseline, Week 104
Population: Participants from the Intent to Treat population who withdrew have been excluded at post withdrawal visits.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 42
Percentage of Participants | 60

23. Secondary Outcome: Part II: Rate of Serious Adverse Events (SAEs), Serious Infection Adverse Events (AEs), Related SAEs, Macrophage Activation Syndrome, AEs Leading to Withdrawal and Deaths Per 100 Patient Years to Week 104
Description: Rate of SAEs, Rate of Serious Infection AEs, Rate of Related SAEs (remotely, possibly, probably) to Tocilizumab (TCZ), Rate of Macrophage Activation Syndrome, Rate of AEs leading to withdrawal and Rate of deaths per 100 patient years (PY) were calculated using the formula:
  Number of Patient Events / Duration in study (years) * 100.
  Multiple occurrences of the same AE in one individual are counted.
Time Frame: 104 Weeks
Population: Safety Population- all participants who received at least one dose of study drug and had 1 post-baseline safety assessment. Includes all safety data in the database up to the week 104 infusion based on the date of randomization for each patient. (Last date was 31 May 2011)
Measure: Number; unit: Events per 100 patient year
Arm/Group | Tocilizumab
Number analyzed (Participants) | 112
Events per 100 patient year
  SAEs | 23.3
  Serious infection AEs | 10.9
  SAEs related to TCZ | 7.4
  Macrophage activation syndrome | 1.5
  AEs leading to withdrawal | 3.0
  Deaths | 1.5

24. Secondary Outcome: Part III: Percentage of Participants With at Least 30%, 50%, 70%, and 90% Improvement in JIA Core Set According to ACR
Description: Percentage of participants with ≥30%, 50%, 70%, and 90% improvement in ACR core set consisting of 6 components: 1) Physician's global assessment of disease activity VAS, 2) Parent/Patient global assessment of overall well-being VAS, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate, and 6) CHAQ-DI consisting of 30 questions in 8 domains.
Time Frame: Weeks 104, 116, 128, 140, 152, 164, 176, 188, 200, 212, 224, 236, 248 and 260
Population: The Part III intent-to-treat (ITT3) population consists of all participants who entered into Part III of the study and received at least one administration of tocilizumab during Part III.
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 42 | 47
percentage of participants
  Week 104 JIA ACR30 (n=42,47) | 100.0 | 100.0
  Week 104 JIA ACR50 (n=42,47) | 100.0 | 100.0
  Week 104 JIA ACR70 (n=42,47) | 92.9 | 95.7
  Week 104 JIA ACR90 (n=42,47) | 81.0 | 72.3
  Week 116 JIA ACR30 (n=41,45) | 100.0 | 100.0
  Week 116 JIA ACR50 (n=41,45) | 100.0 | 97.8
  Week 116 JIA ACR70 (n=41,45) | 95.1 | 97.8
  Week 116 JIA ACR90 (n=41,45) | 82.9 | 80.0
  Week 128 JIA ACR30 (n=39,41) | 100.0 | 100.0
  Week 128 JIA ACR50 (n=39,41) | 100.0 | 100.0
  Week 128 JIA ACR70 (n=39,41) | 97.4 | 97.6
  Week 128 JIA ACR90 (n=39,41) | 79.5 | 82.9
  Week 140 JIA ACR30 (n=34,37) | 100.0 | 100.0
  Week 140 JIA ACR50 (n=34,37) | 100.0 | 100.0
  Week 140 JIA ACR70 (n=34,37) | 100.0 | 94.6
  Week 140 JIA ACR90 (n=34,37) | 73.5 | 75.7
  Week 152 JIA ACR30 (n=27,28) | 100.0 | 100.0
  Week 152 JIA ACR50 (n=27,28) | 100.0 | 100.0
  Week 152 JIA ACR70 (n=27,28) | 100.0 | 96.4
  Week 152 JIA ACR90 (n=27,28) | 66.7 | 78.6
  Week 164 JIA ACR30 (n=27,24) | 100.0 | 100.0
  Week 164 JIA ACR50 (n=27,24) | 100.0 | 100.0
  Week 164 JIA ACR70 (n=27,24) | 92.6 | 95.8
  Week 164 JIA ACR90 (n=27,24) | 66.7 | 75.0
  Week 176 JIA ACR30 (n=22,22) | 100.0 | 100.0
  Week 176 JIA ACR50 (n=22,22) | 100.0 | 100.0
  Week 176 JIA ACR70 (n=22,22) | 100.0 | 95.5
  Week 176 JIA ACR90 (n=22,22) | 63.6 | 63.6
  Week 188 JIA ACR30 (n=20,22) | 100.0 | 100.0
  Week 188 JIA ACR50 (n=20,22) | 100.0 | 100.0
  Week 188 JIA ACR70 (n=20,22) | 95.0 | 95.5
  Week 188 JIA ACR90 (n=20,22) | 45.0 | 72.7
  Week 200 JIA ACR30 (n=19,19) | 100.0 | 100.0
  Week 200 JIA ACR50 (n=19,19) | 100.0 | 94.7
  Week 200 JIA ACR70 (n=19,19) | 94.7 | 89.5
  Week 200 JIA ACR90 (n=19,19) | 63.2 | 78.9
  Week 212 JIA ACR30 (n=18,18) | 100.0 | 100.0
  Week 212 JIA ACR50 (n=18,18) | 100.0 | 94.4
  Week 212 JIA ACR70 (n=18,18) | 100.0 | 94.4
  Week 212 JIA ACR90 (n=18,18) | 72.2 | 77.8
  Week 224 JIA ACR30 (n=17,18) | 100.0 | 100.0
  Week 224 JIA ACR50 (n=17,18) | 100.0 | 88.9
  Week 224 JIA ACR70 (n=17,18) | 100.0 | 88.9
  Week 224 JIA ACR90 (n=17,18) | 64.7 | 83.3
  Week 236 JIA ACR30 (n=16,17) | 100.0 | 100.0
  Week 236 JIA ACR50 (n=16,17) | 100.0 | 100.0
  Week 236 JIA ACR70 (n=16,17) | 93.8 | 100.0
  Week 236 JIA ACR90 (n=16,17) | 68.8 | 88.2
  Week 248 JIA ACR30 (n=15,17) | 100.0 | 100.0
  Week 248 JIA ACR50 (n=15,17) | 100.0 | 100.0
  Week 248 JIA ACR70 (n=15,17) | 86.7 | 94.1
  Week 248 JIA ACR90 (n=15,17) | 73.3 | 70.6
  Week 260 JIA ACR30 (n=15,15) | 100.0 | 93.3
  Week 260 JIA ACR50 (n=15,15) | 93.3 | 93.3
  Week 260 JIA ACR70 (n=15,15) | 86.7 | 93.3
  Week 260 JIA ACR90 (n=15,15) | 60.0 | 66.7

25. Secondary Outcome: Part III: Percentage of Participants Who Maintain JIA ACR30, JIA ACR50, JIA ACR70, JIA ACR90 Response for 6 Months Previous to the Specified Week
Description: JIA ACR core set consisting of 6 components: 1) Physician's global assessment of disease activity VAS, 2) Parent/Patient global assessment of overall well-being VAS, 3) Maximum number of joints with active arthritis, 4) Number of joints with limitation of movement, 5) Erythrocyte Sedimentation Rate, and 6) CHAQ-DI consisting of 30 questions in 8 domains.
Time Frame: Weeks 104, 116, 128, 140, 152, 164, 176, 188, 200, 212, 224, 236, 248 and 260
Population: The Part III ITT3 population
Measure: Number; unit: percentage of participants
Groups:
- All Participants Treated With Tocilizumab: Tocilizumab either 8 mg/kg (participants ≥ 30 kg) or 12 mg/kg (participants <30 kg) iv every 2 weeks for 12 weeks in Part I, every 2 weeks for 92 weeks in Part II and every 2 weeks for 156 weeks in Part III.
  Participants remained on their prescribed standard of care treatment with NSAIDs, methotrexate and corticosteroids if applicable.
Arm/Group | All Participants Treated With Tocilizumab
Number analyzed (Participants) | 89
percentage of participants
  Week 104 JIA ACR 30 (n=89) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 104 JIA ACR 50 (n=89) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 104 JIA ACR 70 (n=89) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 104 JIA ACR 90 (n=89) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 116 JIA ACR 30 (n=86) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 116 JIA ACR 50 (n=86) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 116 JIA ACR 70 (n=86) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 116 JIA ACR 90 (n=86) | NA — Week 104 is the start of Part III. The first 6 month maintenance data starts at Week 128 (24 weeks after Week 104)
  Week 128 JIA ACR 30 (n=80) | 100.0
  Week 128 JIA ACR 50 (n=80) | 98.8
  Week 128 JIA ACR 70 (n=80) | 91.3
  Week 128 JIA ACR 90 (n=80) | 68.8
  Week 140 JIA ACR30 (n=71) | 100.0
  Week 140 JIA ACR50 (n=71) | 98.6
  Week 140 JIA ACR70 (n=71) | 93.0
  Week 140 JIA ACR90 (n=71) | 66.2
  Week 152 JIA ACR30 (n=55) | 100.0
  Week 152 JIA ACR50 (n=55) | 100.0
  Week 152 JIA ACR70 (n=55) | 94.5
  Week 152 JIA ACR90 (n=55) | 60.0
  Week 164 JIA ACR30 (n=51) | 100.0
  Week 164 JIA ACR50 (n=51) | 100.0
  Week 164 JIA ACR70 (n=51) | 92.2
  Week 164 JIA ACR90 (n=51) | 56.9
  Week 176 JIA ACR30 (n=44) | 100.0
  Week 176 JIA ACR50 (n=44) | 100.0
  Week 176 JIA ACR70 (n=44) | 88.6
  Week 176 JIA ACR90 (n=44) | 52.3
  Week 188 JIA ACR30 (n=42) | 100.0
  Week 188 JIA ACR50 (n=42) | 100.0
  Week 188 JIA ACR70 (n=42) | 88.1
  Week 188 JIA ACR90 (n=42) | 50.0
  Week 200 JIA ACR30 (n=38) | 100.0
  Week 200 JIA ACR50 (n=38) | 97.4
  Week 200 JIA ACR70 (n=38) | 86.8
  Week 200 JIA ACR90 (n=38) | 52.6
  Week 212 JIA ACR30 (n=36) | 100.0
  Week 212 JIA ACR50 (n=36) | 97.2
  Week 212 JIA ACR70 (n=36) | 88.9
  Week 212 JIA ACR90 (n=36) | 55.6
  Week 224 JIA ACR30 (n=35) | 100.0
  Week 224 JIA ACR50 (n=35) | 94.3
  Week 224 JIA ACR70 (n=35) | 91.4
  Week 224 JIA ACR90 (n=35) | 68.6
  Week 236 JIA ACR30 (n=33) | 100.0
  Week 236 JIA ACR50 (n=33) | 93.9
  Week 236 JIA ACR70 (n=33) | 90.9
  Week 236 JIA ACR90 (n=33) | 72.7
  Week 248 JIA ACR30 (n=32) | 100.0
  Week 248 JIA ACR50 (n=32) | 93.8
  Week 248 JIA ACR70 (n=32) | 87.5
  Week 248 JIA ACR90 (n=32) | 65.6
  Week 260 JIA ACR30 (n=30) | 96.7
  Week 260 JIA ACR50 (n=30) | 93.3
  Week 260 JIA ACR70 (n=30) | 80.0
  Week 260 JIA ACR90 (n=30) | 56.7

26. Secondary Outcome: Part III: Doses of Oral Corticosteroids
Description: Oral corticosteroid values summarized are based on average daily dose on the nominal study day. The prednisone equivalent is used in calculation of oral corticosteroid dose. Participants who withdrew are excluded at the the visit of withdrawal and all subsequent visits.
Time Frame: Baseline and Weeks 104, 116, 128, 140, 152, 164, 176, 188, 200, 212, 224, 236, 248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 53 | 59
mg/kg/day
  Baseline (n=53,59) | 0.203 (0.1572) | 0.356 (0.1397)
  Week 104 (n=45,48) | 0.020 (0.0455) | 0.047 (0.0869)
  Week 116 (n=42,46) | 0.022 (0.0464) | 0.046 (0.0831)
  Week 128 (n=41,42) | 0.022 (0.0449) | 0.058 (0.1635)
  Week 140 (n=34,38) | 0.031 (0.0625) | 0.051 (0.1112)
  Week 152 (n=28,31) | 0.021 (0.0388) | 0.060 (0.1125)
  Week 164 (n=28,25) | 0.018 (0.0349) | 0.068 (0.1179)
  Week 176 (n=25,23) | 0.019 (0.0383) | 0.073 (0.1327)
  Week 188 (n=21,22) | 0.020 (0.0366) | 0.075 (0.1275)
  Week 200 (n=20,20) | 0.017 (0.0284) | 0.083 (0.1397)
  Week 212 (n=19,19) | 0.016 (0.0274) | 0.077 (0.1449)
  Week 224 (n=18,19) | 0.017 (0.0279) | 0.075 (0.1399)
  Week 236 (n=17,18) | 0.018 (0.0283) | 0.077 (0.1436)
  Week 248 (n=16,18) | 0.020 (0.0290) | 0.076 (0.1429)
  Week 260 (n=16,18) | 0.019 (0.0282) | 0.079 (0.1486)

27. Secondary Outcome: Part III: Percentage of Participants on Corticosteroids at Baseline Able to Discontinue Corticosteroids by Weeks 104,116, 128, 140, 152, 164, 176, 188, 200, 212, 224, 236, 248, and 260
Description: Values summarized are based on average daily dose on the nominal study day. The prednisone equivalent is used in calculation of oral corticosteroid dose. Participants who withdrew are excluded at the timepoint of this event and at all subsequent visits.
  Baseline considered first dose of study treatment. Data presented up to entry into the Alternative Dosing Schedule.
Time Frame: Weeks 104,116, 128, 140, 152, 164, 176, 188, 200, 212, 224, 236, 248, and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 38 | 46
percentage of participants
  Week 104 (n=38,46) | 66.0 | 67.0
  Week 116 (n=36,44) | 67.0 | 68.0
  Week 128 (n=35,40) | 69.0 | 70.0
  Week 140 (n=31,36) | 68 | 67
  Week 152 (n=25,30) | 64.0 | 57.0
  Week 164 (n=25,24) | 68.0 | 58.0
  Week 176 (n=22,22) | 68.0 | 64.0
  Week 188 (n=18,21) | 61.0 | 57.0
  Week 200 (n=17,20) | 59.0 | 60.0
  Week 212 (n=16,19) | 56.0 | 63.0
  Week 224 (n=15,19) | 53.0 | 63.0
  Week 236 (n=14,18) | 50.0 | 61.0
  Week 248 (n=13,18) | 46.0 | 61.0
  Week 260 (n=13,18) | 46.0 | 61.0

28. Secondary Outcome: Part III: Percentage of Participants With a >=20/50/75/90% Decrease From Baseline in Oral Corticosteroid Dose at Visits
Description: Values summarized are based on average daily dose on the nominal study day. The prednisone equivalent is used in calculation of oral corticosteroid dose. Participants who withdrew are excluded at the timepoint of this event and at all subsequent visits.
  Baseline considered first dose of study treatment.
Time Frame: Every 2 weeks from Week 104 to Week 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 38 | 46
percentage of participants
  Week 104 >20% decrease (n=38,46) | 100.0 | 97.8
  Week 104 >50% decrease (n=38,46) | 94.7 | 91.3
  Week 104 >75% decrease (n=38,46) | 84.2 | 82.6
  Week 104 >90% decrease (n=38,46) | 71.1 | 71.7
  Week 106 >20% decrease (n=37,46) | 100.0 | 97.8
  Week 106 >50% decrease (n=37,46) | 91.9 | 91.3
  Week 106 >75% decrease (n=37,46) | 83.8 | 82.6
  Week 106 >90% decrease (n=37,46) | 70.3 | 71.7
  Week 108 >20% decrease (n=37,45) | 100.0 | 100.0
  Week 108 >50% decrease (n=37,45) | 89.2 | 91.1
  Week 108 >75% decrease (n=37,45) | 81.1 | 84.4
  Week 108 >90% decrease (n=37,45) | 70.3 | 73.3
  Week 110 >20% decrease (n=36,44) | 100.0 | 100.0
  Week 110 >50% decrease (n=36,44) | 88.9 | 93.2
  Week 110 >75% decrease (n=36,44) | 80.6 | 84.1
  Week 110 >90% decrease (n=36,44) | 72.2 | 75.0
  Week 112 >20% decrease (n=36,44) | 100.0 | 100.0
  Week 112 >50% decrease (n=36,44) | 88.9 | 95.5
  Week 112 >75% decrease (n=36,44) | 80.6 | 81.8
  Week 112 >90% decrease (n=36,44) | 72.2 | 75.0
  Week 114 >20% decrease (n=36,44) | 100.0 | 100.0
  Week 114 >50% decrease (n=36,44) | 88.9 | 95.5
  Week 114 >75% decrease (n=36,44) | 80.6 | 79.5
  Week 114 >90% decrease (n=36,44) | 72.2 | 72.7
  Week 116 >20% decrease (n=35,44) | 100.0 | 100.0
  Week 116 >50% decrease (n=35,44) | 91.4 | 93.2
  Week 116 >75% decrease (n=35,44) | 80.0 | 79.5
  Week 116 >90% decrease (n=35,44) | 71.4 | 72.7
  Week 118 >20% decrease (n=35,43) | 100.0 | 100.0
  Week 118 >50% decrease (n=35,43) | 88.6 | 93.0
  Week 118 >75% decrease (n=35,43) | 80.0 | 81.4
  Week 118 >90% decrease (n=35,43) | 71.4 | 74.4
  Week 120 >20% decrease (n=35,43) | 100.0 | 100.0
  Week 120 >50% decrease (n=35,43) | 88.6 | 93.0
  Week 120 >75% decrease (n=35,43) | 80.0 | 83.7
  Week 120 >90% decrease (n=35,43) | 74.3 | 76.7
  Week 122 >20% decrease (n=35,43) | 97.1 | 100.0
  Week 122 >50% decrease (n=35,43) | 88.6 | 93.0
  Week 122>75% decrease (n=35,43) | 77.1 | 81.4
  Week 122 >90% decrease (n=35,43) | 74.3 | 74.4
  Week 124 >20% decrease (n=35,43) | 100.0 | 100.0
  Week 124 >50% decrease (n=35,43) | 94.3 | 93.0
  Week 124 >75% decrease (n=35,43) | 80.0 | 83.7
  Week 124 >90% decrease (n=35,43) | 77.1 | 74.4
  Week 126 >20% decrease (n=35,43) | 100.0 | 100.0
  Week 126 >50% decrease (n=35,43) | 94.3 | 90.7
  Week 126 >75% decrease (n=35,43) | 80.0 | 81.4
  Week 126 >90% decrease (n=35,43) | 77.1 | 74.4
  Week 128 >20% decrease (n=35,39) | 100.0 | 97.4
  Week 128 >50% decrease (n=35,39) | 91.4 | 89.7
  Week 128 >75% decrease (n=35,39) | 80.0 | 82.1
  Week 128 >90% decrease (n=35,39) | 77.1 | 71.8
  Week 130 >20% decrease (n=35,39) | 100.0 | 97.4
  Week 130 >50% decrease (n=35,39) | 91.4 | 89.7
  Week 130 >75% decrease (n=35,39) | 80.0 | 87.2
  Week 130 >90% decrease (n=35,39) | 80.0 | 74.4
  Week 132 >20% decrease (n=35,39) | 100.0 | 97.4
  Week 132 >50% decrease (n=35,39) | 91.4 | 87.2
  Week 132 >75% decrease (n=35,39) | 80.0 | 84.6
  Week 132 >90% decrease (n=35,39) | 80.0 | 71.8
  Week 134 >20% decrease (n=35,39) | 94.3 | 97.4
  Week 134 >50% decrease (n=35,39) | 88.6 | 87.2
  Week 134 >75% decrease (n=35,39) | 77.1 | 84.6
  Week 134 >90% decrease (n=35,39) | 77.1 | 71.8
  Week 136 >20% decrease (n=34,39) | 97.1 | 97.4
  Week 136 >50% decrease (n=34,39) | 91.2 | 89.7
  Week 136 >75% decrease (n=34,39) | 76.5 | 84.6
  Week 136 >90% decrease (n=34,39) | 76.5 | 71.8
  Week 138 >20% decrease (n=34,39) | 94.1 | 97.4
  Week 138 >50% decrease (n=34,39) | 88.2 | 89.7
  Week 138 >75% decrease (n=34,39) | 76.5 | 84.6
  Week 138 >90% decrease (n=34,39) | 76.5 | 71.8
  Week 140 >20% decrease (n=29,36) | 93.1 | 97.2
  Week 140 >50% decrease (n=29,36) | 86.2 | 88.9
  Week 140 >75% decrease (n=29,36) | 72.4 | 83.3
  Week 140 >90% decrease (n=29,36) | 72.4 | 72.2
  Week 142 >20% decrease (n=29,36) | 93.1 | 97.2
  Week 142 >50% decrease (n=29,36) | 86.2 | 88.9
  Week 142 >75% decrease (n=29,36) | 72.4 | 83.3
  Week 142 >90% decrease (n=29,36) | 69.0 | 72.2
  Week 144 >20% decrease (n=28,36) | 92.9 | 97.2
  Week 144 >50% decrease (n=28,36) | 89.3 | 88.9
  Week 144 >75% decrease (n=28,36) | 71.4 | 83.3
  Week 144 >90% decrease (n=28,36) | 67.9 | 72.2
  Week 146 >20% decrease (n=28,36) | 96.4 | 97.2
  Week 146 >50% decrease (n=28,36) | 92.9 | 86.1
  Week 146 >75% decrease (n=28,36) | 75.0 | 80.6
  Week 146 >90% decrease (n=28,36) | 71.4 | 66.7
  Week 148 >20% decrease (n=27,35) | 100.0 | 97.1
  Week 148 >50% decrease (n=27,35) | 96.3 | 85.7
  Week 148 >75% decrease (n=27,35) | 77.8 | 80.0
  Week 148 >90% decrease (n=27,35) | 74.1 | 65.7
  Week 150 >20% decrease (n=25,35) | 100.0 | 97.1
  Week 150 >50% decrease (n=25,35) | 96.0 | 88.6
  Week 150 >75% decrease (n=25,35) | 76.0 | 80.0
  Week 150 >90% decrease (n=25,35) | 76.0 | 68.6
  Week 152 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 152 >50% decrease (n=25,27) | 96.0 | 85.2
  Week 152 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 152 >90% decrease (n=25,27) | 76.0 | 63.0
  Week 154 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 154 >50% decrease (n=25,27) | 96.0 | 88.9
  Week 154 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 154 >90% decrease (n=25,27) | 76.0 | 70.4
  Week 156 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 156 >50% decrease (n=25,27) | 96.0 | 85.2
  Week 156 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 156 >90% decrease (n=25,27) | 76.0 | 70.4
  Week 158 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 158 >50% decrease (n=25,27) | 96.0 | 88.9
  Week 158 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 158 >90% decrease (n=25,27) | 76.0 | 70.4
  Week 160 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 160 >50% decrease (n=25,27) | 96.0 | 85.2
  Week 160 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 160 >90% decrease (n=25,27) | 76.0 | 70.4
  Week 162 >20% decrease (n=25,27) | 100.0 | 96.3
  Week 162 >50% decrease (n=25,27) | 96.0 | 81.5
  Week 162 >75% decrease (n=25,27) | 76.0 | 77.8
  Week 162 >90% decrease (n=25,27) | 76.0 | 70.4
  Week 164 >20% decrease (n=24,24) | 100.0 | 95.8
  Week 164 >50% decrease (n=24,24) | 95.8 | 83.3
  Week 164 >75% decrease (n=24,24) | 75.0 | 75.0
  Week 164 >90% decrease (n=24,24) | 75.0 | 70.8
  Week 166 >20% decrease (n=24,22) | 100.0 | 95.5
  Week 166 >50% decrease (n=24,22) | 95.8 | 81.8
  Week 166 >75% decrease (n=24,22) | 75.0 | 72.7
  Week 166 >90% decrease (n=24,22) | 75.0 | 68.2
  Week 168 >20% decrease (n=24,22) | 100.0 | 95.5
  Week 168 >50% decrease (n=24,22) | 95.8 | 81.8
  Week 168 >75% decrease (n=24,22) | 75.0 | 72.7
  Week 168 >90% decrease (n=24,22) | 75.0 | 68.2
  Week 170 >20% decrease (n=22,22) | 100.0 | 90.9
  Week 170 >50% decrease (n=22,22) | 95.5 | 81.8
  Week 170 >75% decrease (n=22,22) | 77.3 | 72.7
  Week 170 >90% decrease (n=22,22) | 77.3 | 68.2
  Week 172 >20% decrease (n=22,22) | 100.0 | 90.9
  Week 172 >50% decrease (n=22,22) | 95.5 | 90.9
  Week 172 >75% decrease (n=22,22) | 77.3 | 72.7
  Week 172 >90% decrease (n=22,22) | 77.3 | 68.2
  Week 174 >20% decrease (n=22,22) | 100.0 | 90.9
  Week 174 >50% decrease (n=22,22) | 95.5 | 90.9
  Week 174 >75% decrease (n=22,22) | 77.3 | 72.7
  Week 174 >90% decrease (n=22,22) | 77.3 | 68.2
  Week 176 >20% decrease (n=19,22) | 100.0 | 90.9
  Week 176 >50% decrease (n=19,22) | 94.7 | 90.9
  Week 176 >75% decrease (n=19,22) | 73.7 | 72.7
  Week 176 >90% decrease (n=19,22) | 73.7 | 68.2
  Week 178 >20% decrease (n=19,22) | 100.0 | 90.9
  Week 178 >50% decrease (n=19,22) | 94.7 | 90.9
  Week 178 >75% decrease (n=19,22) | 73.7 | 72.7
  Week 178 >90% decrease (n=19,22) | 73.7 | 68.2
  Week 180 >20% decrease (n=19,22) | 100.0 | 90.9
  Week 180 >50% decrease (n=19,22) | 94.7 | 90.9
  Week 180 >75% decrease (n=19,22) | 73.7 | 68.2
  Week 180 >90% decrease (n=19,22) | 73.7 | 63.6
  Week 182 >20% decrease (n=18,22) | 100.0 | 90.9
  Week 182 >50% decrease (n=18,22) | 94.4 | 90.9
  Week 182 >75% decrease (n=18,22) | 72.2 | 68.2
  Week 182 >90% decrease (n=18,22) | 72.2 | 63.6
  Week 184 >20% decrease (n=18,22) | 100.0 | 90.9
  Week 184 >50% decrease (n=18,22) | 94.4 | 86.4
  Week 184 >75% decrease (n=18,22) | 72.2 | 68.2
  Week 184 >90% decrease (n=18,22) | 72.2 | 63.6
  Week 186 >20% decrease (n=18,22) | 100.0 | 90.0
  Week 186 >50% decrease (n=18,22) | 94.4 | 90.9
  Week 186 >75% decrease (n=18,22) | 72.2 | 68.2
  Week 186 >90% decrease (n=18,22) | 72.2 | 63.6
  Week 188 >20% decrease (n=18,21) | 100.0 | 90.5
  Week 188 >50% decrease (n=18,21) | 94.4 | 90.5
  Week 188 >75% decrease (n=18,21) | 72.2 | 71.4
  Week 188 >90% decrease (n=18,21) | 72.2 | 61.9
  Week 190 >20% decrease (n=18,21) | 100.0 | 95.2
  Week 190 >50% decrease (n=18,21) | 94.4 | 85.7
  Week 190 >75% decrease (n=18,21) | 72.2 | 66.7
  Week 190 >90% decrease (n=18,21) | 72.2 | 61.9
  Week 192 >20% decrease (n=18,21) | 100.0 | 95.2
  Week 192 >50% decrease (n=18,21) | 94.4 | 81.0
  Week 192 >75% decrease (n=18,21) | 72.2 | 66.7
  Week 192 >90% decrease (n=18,21) | 72.2 | 61.9
  Week 194 >20% decrease (n=18,20) | 100.0 | 95.0
  Week 194 >50% decrease (n=18,20) | 94.4 | 80.0
  Week 194 >75% decrease (n=18,20) | 72.2 | 70.0
  Week 194 >90% decrease (n=18,20) | 72.2 | 65.0
  Week 196 >20% decrease (n=18,20) | 100.0 | 90.0
  Week 196 >50% decrease (n=18,20) | 94.4 | 80.0
  Week 196 >75% decrease (n=18,20) | 72.2 | 70.0
  Week 196 >90% decrease (n=18,20) | 72.2 | 65.0
  Week 198 >20% decrease (n=18,20) | 100.0 | 90.0
  Week 198 >50% decrease (n=18,20) | 94.4 | 80.0
  Week 198 >75% decrease (n=18,20) | 72.2 | 70.0
  Week 198 >90% decrease (n=18,20) | 72.2 | 65.0
  Week 200 >20% decrease (n=17,20) | 100.0 | 90.0
  Week 200 >50% decrease (n=17,20) | 94.1 | 85.0
  Week 200 >75% decrease (n=17,20) | 76.5 | 75.0
  Week 200 >90% decrease (n=17,20) | 70.6 | 65.0
  Week 202 >20% decrease (n=17,20) | 100.0 | 90.0
  Week 202 >50% decrease (n=17,20) | 94.1 | 85.0
  Week 202 >75% decrease (n=17,20) | 76.5 | 75.0
  Week 202 >90% decrease (n=17,20) | 70.6 | 65.0
  Week 204 >20% decrease (n=17,20) | 100.0 | 90.0
  Week 204 >50% decrease (n=17,20) | 94.1 | 85.0
  Week 204 >70% decrease (n=17,20) | 76.5 | 75.0
  Week 204 >90% decrease (n=17,20) | 70.6 | 65.0
  Week 206 >20% decrease (n=16,20) | 100.0 | 85.0
  Week 206 >50% decrease (n=16,20) | 93.8 | 75.0
  Week 206 >75% decrease (n=16,20) | 75.0 | 75.0
  Week 206 >90% decrease (n=16,20) | 68.8 | 70.0
  Week 208 >20% decrease (n=16,20) | 100.0 | 90.0
  Week 208 >50% decrease (n=16,20) | 93.8 | 80.0
  Week 208 >75% decrease (n=16,20) | 75.0 | 75.0
  Week 208 >90% decrease (n=16,20) | 68.8 | 70.0
  Week 210 >20% decrease (n=16,19) | 100.0 | 89.5
  Week 210 >50% decrease (n=16,19) | 93.8 | 84.2
  Week 210 >75% decrease (n=16,19) | 81.3 | 78.9
  Week 210 >90% decrease (n=16,19) | 75.0 | 73.7
  Week 212 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 212 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 212 >75% decrease (n=15,19) | 73.3 | 78.9
  Week 212 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 214 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 214 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 214 >75% decrease (n=15,19) | 73.3 | 78.9
  Week 214 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 216 >20% decrease (n=15,19) | 100.0 | 94.7
  Week 216 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 216 >75% decrease (n=15,19) | 73.3 | 78.9
  Week 216 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 218 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 218 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 218 >75% decrease (n=15,19) | 80.0 | 78.9
  Week 218 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 220 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 220 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 220 >75% decrease (n=15,19) | 80.0 | 78.9
  Week 220 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 222 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 222 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 222 >75% decrease (n=15,19) | 80.0 | 78.9
  Week 222 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 224 >20% decrease (n=15,19) | 100.0 | 89.5
  Week 224 >50% decrease (n=15,19) | 93.3 | 84.2
  Week 224 >75% decrease (n=15,19) | 80.0 | 78.9
  Week 224 >90% decrease (n=15,19) | 73.3 | 73.7
  Week 226 >20% decrease (n=14,19) | 100.0 | 89.5
  Week 226 >50% decrease (n=14,19) | 92.9 | 84.2
  Week 226 >75% decrease (n=14,19) | 78.6 | 78.9
  Week 226 >90% decrease (n=14,19) | 71.4 | 73.7
  Week 228 >20% decrease (n=14,19) | 100.0 | 89.5
  Week 228 >50% decrease (n=14,19) | 92.9 | 89.5
  Week 228 >75% decrease (n=14,19) | 78.6 | 78.9
  Week 228 >90% decrease (n=14,19) | 71.4 | 73.7
  Week 230 >20% decrease (n=14,19) | 100.0 | 89.5
  Week 230 >50% decrease (n=14,19) | 92.9 | 89.5
  Week 230 >75% decrease (n=14,19) | 78.6 | 78.9
  Week 230 >90% decrease (n=14,19) | 71.4 | 73.7
  Week 232 >20% decrease (n=14,18) | 100.0 | 88.9
  Week 232 >50% decrease (n=14,18) | 92.9 | 88.9
  Week 232 >75% decrease (n=14,18) | 78.6 | 77.8
  Week 232 >90% decrease (n=14,18) | 71.4 | 72.2
  Week 234 >20% decrease (n=14,18) | 100.0 | 88.9
  Week 234 >50% decrease (n=14,18) | 92.9 | 88.9
  Week 234 >75% decrease (n=14,18) | 78.6 | 77.8
  Week 234 >90% decrease (n=14,18) | 71.4 | 72.2
  Week 236 >20% decrease (n=14,18) | 100.0 | 94.4
  Week 236 >50% decrease (n=14,18) | 92.9 | 88.9
  Week 236 >75% decrease (n=14,18) | 78.6 | 77.8
  Week 236 >90% decrease (n=14,18) | 71.4 | 72.2
  Week 238 >20% decrease (n=14,18) | 100.0 | 94.4
  Week 238 >50% decrease (n=14,18) | 92.9 | 88.9
  Week 238 >75% decrease (n=14,18) | 78.6 | 77.8
  Week 238 >90% decrease (n=14,18) | 71.4 | 72.2
  Week 240 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 240 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 240 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 240 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 242 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 242 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 242 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 242 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 244 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 244 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 244 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 244 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 246 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 246 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 246 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 246 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 248 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 248 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 248 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 248 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 250 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 250 >50% decrease (n=13,18) | 92.3 | 83.3
  Week 250 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 250 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 252 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 252 >50% decrease (n=13,18) | 92.3 | 83.3
  Week 252 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 252 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 254 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 254 >50% decrease (n=13,18) | 92.3 | 83.3
  Week 254 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 254 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 256 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 256 >50% decrease (n=13,18) | 92.3 | 83.3
  Week 256 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 256 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 258 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 258 >50% decrease (n=13,18) | 92.3 | 83.3
  Week 258 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 258 >90% decrease (n=13,18) | 69.2 | 72.2
  Week 260 >20% decrease (n=13,18) | 100.0 | 94.4
  Week 260 >50% decrease (n=13,18) | 92.3 | 88.9
  Week 260 >75% decrease (n=13,18) | 76.9 | 77.8
  Week 260 >90% decrease (n=13,18) | 69.2 | 72.2

29. Secondary Outcome: Part III: Percentage of Participants With Inactive Disease
Description: Participants who previously withdrew are excluded.
  Responders are participants who met all of the following criteria for inactive disease at the visit assessment day:
  i. Number of active joints = 0. ii. Absence of lymphadenopathy, hepatomegaly or splenomegaly in the nearest non-missing physical examination prior to or after the week assessment day. This could include results outside of the time window.
  iii. Absence of symptomatic serositis adverse event. iv. In the 14 days preceding the week assessment day no fever (temperature >=37.5 C) or rash characteristic of sJIA.
  v. Normal ESR as defined by an ESR <20 mm/hr regardless of age and sex. vi. Physician global assessment VAS <=10. LOCF rule applied to missing number of active joints, ESR and Physician global assessment VAS.
  Data presented up to the point of entry into the Alternative Dosing Schedule.
Time Frame: Weeks 104, 116, 128, 140, 152, 164, 188, 200, 212, 224,236,248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 42 | 47
percentage of participants
  Week 104 (n=42,47) | 45.2 | 46.8
  Week 116 (n=41,46) | 48.8 | 43.5
  Week 128 (n=40,43) | 55.0 | 48.8
  Week 140 (n=38,40) | 55.3 | 45.0
  Week 152 (n=27,35) | 33.3 | 54.3
  Week 164 (n=27,25) | 37.0 | 28.0
  Week 176 (n=24,22) | 41.7 | 36.4
  Week 188 (n=21,22) | 23.8 | 31.8
  Week 200 (n=19,21) | 42.1 | 14.3
  Week 212 (n=18,18 | 55.6 | 44.4
  Week 224 (n=17,18) | 47.1 | 44.4
  Week 236 (n=16,17) | 43.8 | 29.4
  Week 248 (n=15,17) | 26.7 | 41.2
  Week 260 (n=15,15) | 46.7 | 6.7

30. Secondary Outcome: Part III: Percentage of Participants in Clinical Remission
Description: Patients who previously withdrew are excluded Responders are patients who met all of the following criteria for inactive disease at all visits in the 6 months (180 days) prior to and including the visit assessment day: i. Number of active joints = 0. ii. Absence of lymphadenopathy, hepatomegaly or splenomegaly in the nearest non-missing physical examination prior to or after the week assessment day. This could include results outside of the time window.
  iii. Absence of symptomatic serositis adverse event. iv. In the 14 days preceding the week assessment day no fever (temperature >=37.5 C) or rash characteristic of sJIA. v. Normal ESR as defined by an ESR <20 mm/hr regardless of age and sex.
  vi. iv. Physician global assessment VAS <=10. LOCF rule applied to missing number of active joints, ESR and Physician global assessment VAS. ESR = Erythrocyte Sedimentation Rate. VAS = Visual Analogue Scale. Data presented up to the point of entry into the Alternative Dosing Schedule.
Time Frame: Weeks 116, 128, 140, 152, 164, 188, 200, 212, 224,236,248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 41 | 47
percentage of participants
  Week 116 (n=41,47) | 14.6 | 17.4
  Week 128 (n=40,43) | 32.5 | 23.3
  Week 140 (n=38,40) | 34.2 | 25.0
  Week 152 (n=27,35) | 25.9 | 25.7
  Week 164 (n=27,25) | 22.2 | 16.0
  Week 176 (n=24,22) | 16.7 | 13.6
  Week 188 (n=21,22) | 14.3 | 9.1
  Week 200 (n=19,21) | 15.8 | 4.8
  Week 212 (n=18,18) | 16.7 | 5.6
  Week 224 (n=17,18) | 29.4 | 11.1
  Week 236 (n=16,17) | 25.0 | 29.4
  Week 248 (n=15,17) | 13.3 | 23.5
  Week 260 (n=15,15) | 13.3 | 6.7

31. Secondary Outcome: Part III: Percentage of Participants on Corticosteroids at Baseline in Clinical Remission Off All Oral Corticosteroids for 6 Months Prior to Specified Visits
Description: There were 4 levels of clinical remission defined while the patient remained on tocilizumab as defined below.. After level 1, each successive level required that all the previous level criteria be met:
  Level 1: inactive disease criteria have been met at all assessments in the last 6 months (180 days) preceding the timepoint assessment day Level 2: level 1 criteria and no oral corticosteroids received in the last 6 months (180 days) preceding the timepoint assessment day Level 3: level 2 criteria and no methotrexate received in the last 6 months (180 days) preceding the timepoint assessment day Level 4: level 3 criteria and no NSAIDs received for sJIA in the last 6 months (180 days) preceding the timepoint assessment day
Time Frame: Weeks 116, 128, 140, 152, 164, 188, 200, 212, 224,236,248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 41 | 46
percentage of participants
  Week 116 (n=41,46) | 12.2 | 17.4
  Week 128 (n=40,43) | 32.5 | 20.9
  Week 140 (n=38,40) | 28.9 | 20.0
  Week 152 (n=27,35) | 18.5 | 20.0
  Week 164 (n=27,25) | 18.5 | 12.0
  Week 176 (n=24,22) | 16.7 | 9.1
  Week 188 (n=21,22) | 14.3 | 4.5
  Week 200 (n=19,21) | 10.5 | 4.8
  Week 212 (n=18,18) | 11.1 | 5.6
  Week 224 (n=17,18) | 23.5 | 11.1
  Week 236 (n=16,17) | 25.0 | 23.5
  Week 248 (n=15,17) | 6.7 | 17.6
  Week 260 (n=15,15) | 6.7 | 6.7

32. Secondary Outcome: Part III: Percentage of Participants on Methotrexate At Baseline in Clinical Remission Off Corticosteroids and Methotrexate for 6 Months Prior to Specified Visits
Description: as for outcome 31
Time Frame: Weeks 116, 128, 140, 152, 164, 188, 200, 212, 224,236,248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 41 | 46
percentage of participants
  Week 116 (n=41,46) | 7.3 | 8.7
  Week 128 (n=40,43) | 20.0 | 11.6
  Week 140 (n=38,40) | 18.4 | 5.0
  Week 152 (n=27,35) | 3.7 | 2.9
  Week 164 (n=27,25) | 3.7 | 4.0
  Week 176 (n=24,22) | 4.2 | 0.0
  Week 188 (n=21,22) | 4.8 | 0.0
  Week 200 (n=19,21) | 5.3 | 4.8
  Week 212 (n=18,18) | 5.6 | 5.6
  Week 224 (n=17,18) | 5.9 | 5.6
  Week 236 (n=16,17) | 12.5 | 5.9
  Week 248 (n=15,17) | 0.0 | 5.9
  Week 260 (n=15,15) | 0.0 | 0.0

33. Secondary Outcome: Part III: Percentage of Participants in Clinical Remission Off All Arthritis Medications Except Tocilizumab for 6 Months Prior to Specified Visits
Description: as for outcome 31
Time Frame: Weeks 116, 128, 140, 152, 164, 188, 200, 212, 224,236,248 and 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 41 | 46
percentage of participants
  Week 116 (n=41,46) | 4.9 | 8.7
  Week 128 (n=40,43) | 15.0 | 9.3
  Week 140 (n=38,40) | 15.8 | 5.0
  Week 152 (n=27,35) | 0.0 | 2.9
  Week 164 (n=27,25) | 0.0 | 0.0
  Week 176 (n=24,22) | 4.2 | 0.0
  Week 188 (n=21,22) | 4.8 | 0.0
  Week 200 (n=19,21) | 5.3 | 0.0
  Week 212 (n=18,18) | 5.6 | 0.0
  Week 224 (n=17,18) | 5.9 | 0.0
  Week 236 (n=16,17) | 12.5 | 0.0
  Week 248 (n=15,17) | 0.0 | 0.0
  Week 260 (n=15,15) | 0.0 | 0.0

34. Secondary Outcome: Part III: Percentage of Participants Who Developed Antibodies To Tocilizumab During Weeks 104 to 260
Description: Human antibodies against human antibodies (HAHA), anti-tocilizumab antibodies were assessed by immunogenicity techniques from blood samples drawn every two weeks during Part III of the study.
Time Frame: Every 2 weeks from Week 104 to 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 45 | 47
percentage of participants | 0.0 | 0.0

35. Secondary Outcome: Part III: Percentage of Participants Who Developed Anti-TCZ Antibodies Associated With The Occurrence of Drug Hypersensitivity Reactions.
Description: as for outcome 34
Time Frame: Every 2 weeks from Week 104 to 260
Population: ITT3 population; n=number of participants contributing to the specific statistic
Measure: Number; unit: percentage of participants
Arm/Group | Participants ≥30 kg | Participants <30 kg
Number analyzed (Participants) | 45 | 47
percentage of participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: AE onset between time of very first drug intake and date of last contact or 30 days after very last drug intake. 30 days after 12 weeks of treatment in Part I, 30 days after up to Week 104 in Part II and 30 days after up to Week 260 in Part III .
Description: Note: Adverse Events (AEs) reported in the All Tocilizumab (Part I, Part II and Part III) arm are cumulative to Week 260 and include AEs previously reported in the Tocilizumab_8 mg/kg (Part I) and Tocilizumab_12 mg/kg (Part I) arms that occurred in the 12 week treatment period.
Groups:
- All Tocilizumab (Part I, Part II and Part III): Tocilizumab either 8 mg/kg (participants ≥ 30 kg) or 12 mg/kg (participants <30 kg) iv every 2 weeks for 12 weeks in Part I, every 2 weeks for 92 weeks in Part II and every 2 weeks for 156 weeks in Part III.
Arm/Group | All Tocilizumab (Part I, Part II and Part III)
Serious Adverse Events (participants affected / at risk) | 48/112
Other Adverse Events (participants affected / at risk) | 112/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Tocilizumab (Part I, Part II and Part III) (N=112)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 5
Lymphadenitis (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Drug intolerance (General disorders) | 1
Influenza like illness (General disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Kidney infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pulmonary tuberculosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 5
Femur fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Acute Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Self injurious behavior (Psychiatric disorders) | 1
Testicular torsion (Reproductive system and breast disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.68% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Tocilizumab (Part I, Part II and Part III) (N=112)
Upper Respiratory Tract Infection (Infections and infestations) | 49
Nasopharyngitis (Infections and infestations) | 53
Gastroenteritis viral (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 20
Pyrexia (General disorders) | 11
Influenza like illness (General disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 29
Abdominal pain (Gastrointestinal disorders) | 16
Gastrointestinal disorder (Gastrointestinal disorders) | 6
Haematuria (Renal and urinary disorders) | 5
Dysmenorrhoea (Reproductive system and breast disorders) | 3
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 12
Headache (Nervous system disorders) | 25
Dizziness (Nervous system disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 45
Urticaria (Skin and subcutaneous tissue disorders) | 8
Gastroenteritis (Infections and infestations) | 28
Ear infection (Infections and infestations) | 18
Rhinitis (Infections and infestations) | 19
Impetigo (Infections and infestations) | 14
Viral infection (Infections and infestations) | 16
Otitis media (Infections and infestations) | 14
Viral upper respiratory tract infection (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 11
Otitis externa (Infections and infestations) | 8
Tonsillitis (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 10
Nausea (Gastrointestinal disorders) | 26
Abdominal pain upper (Gastrointestinal disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 9
Contusion (Injury, poisoning and procedural complications) | 10
Excoriation (Injury, poisoning and procedural complications) | 8
Joint injury (Injury, poisoning and procedural complications) | 7
Traumatic haematoma (Injury, poisoning and procedural complications) | 7
Rash (Skin and subcutaneous tissue disorders) | 22
Eczema (Skin and subcutaneous tissue disorders) | 10
Prurigo (Skin and subcutaneous tissue disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 11
Transaminases increased (Investigations) | 11
Conjunctivitis (Infections and infestations) | 12
Haematoma (Vascular disorders) | 7
Sinusitis (Infections and infestations) | 10
Influenza (Infections and infestations) | 9
Paronychia (Infections and infestations) | 7
Herpes Zoster (Infections and infestations) | 6
Laryngitis (Infections and infestations) | 6
Dental Caries (Gastrointestinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Joint Swelling (Musculoskeletal and connective tissue disorders) | 7
Ligament Sprain (Injury, poisoning and procedural complications) | 13
Limb Injury (Injury, poisoning and procedural complications) | 8
Fall (Injury, poisoning and procedural complications) | 7
Wound (Injury, poisoning and procedural complications) | 6
Lymphadenopathy (Blood and lymphatic system disorders) | 6
Fatigue (General disorders) | 6
Arthropod bite (Injury, poisoning and procedural complications) | 17
Local swelling (General disorders) | 5
Pain (General disorders) | 4
Hand fracture (Injury, poisoning and procedural complications) | 5
Laceration (Injury, poisoning and procedural complications) | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Muscle strain (Injury, poisoning and procedural complications) | 4
Thermal burn (Injury, poisoning and procedural complications) | 4
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 4
Lymphadenitis (Blood and lymphatic system disorders) | 4
Migraine (Nervous system disorders) | 3
Cataract (Eye disorders) | 4
Chalazion (Eye disorders) | 3
Ear pain (Ear and labyrinth disorders) | 11
Middle ear effusion (Ear and labyrinth disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Cellulitis (Infections and infestations) | 5
Skin infection (Infections and infestations) | 5
Tinea pedis (Infections and infestations) | 5
Varicella (Infections and infestations) | 4
Otitis media acute (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 3

LIMITATIONS AND CAVEATS:
This study consists of 3 parts:

Part I: a 12 week double-blind placebo controlled study is complete. Part II: a 92 week single arm open-label extension study- CSR completed Dec. 2011.

Part III: a 3 year open label continuation study is ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.